CLINICAL TRIAL: NCT05206864
Title: Food Trial to Evaluate the Safety and Tolerability of SBD111 in Health Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solarea Bio, Inc (Industry)
Collaborators: Hebrew SeniorLife (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Pro00054643
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBD111 (Experimental)
  Interventions: Other: Medical Food: SBD111
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Medical Food: SBD111 — One capsule administered twice daily with morning and evening meals for 28 days
  Arms: SBD111
Other: Placebo — One capsule administered twice daily with morning and evening meals for 28 days
  Arms: Placebo

SUMMARY:
The aim of the trial is to determine if the synbiotic (prebiotic and probiotic), provided twice daily (capsule) is safe and tolerable in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Stated availability throughout entire study period and willingness to fulfill all details of the protocol
3. Age 18-70
4. Be in general good health as determined by a screening evaluation within 30 days of the first dose of SBD111 or placebo
5. Willing to comply with protocol and report on compliance and side effects during study period
6. Body Mass Index between 18.5 and 35 kg/m2
7. Normal cardiovascular parameters, systolic blood pressure ≤ 155 mm Hg, diastolic blood pressure ≤ 95 mm Hg)

Exclusion Criteria:

1. Are currently taking probiotic or prebiotic supplements, or have taken them in the past 30 days
2. Unwilling to avoid probiotics/prebiotics supplements for the duration of the study
3. Known or suspected allergies to probiotics
4. Received oral or parenteral antibiotics within 3 months of enrollment or prescribed antibiotics on day of enrollment.
5. Major surgery or endoscopy within last 3 months.
6. Subject is a smoker
7. Subject has a history of drug and/or alcohol abuse at the time of enrolment
8. Presence of any of the following:
9. Abnormal vital signs or clinically significant systems abnormalities based on screening questionnaire
10. Indwelling catheter or implanted hardware/prosthetic device or feeding tube
11. Febrile illness (oral temperature >37 degrees Celsius) or one or more episodes of diarrhea within 72 hours of baseline visit (first dose of study drug)
12. Active bowel leak, acute abdomen, colitis, or active GI disease or history of gastric or intestinal dysmotility, slowed transit time, variable small intestinal permeability, pancreatitis, or inflammatory bowel disease
13. History of Hepatitis B or Hepatitis C infections, cirrhosis, or chronic liver disease
14. Underlying structural heart disease or previous history of endocarditis or valve replacement
15. Immunosuppression including HIV positive, solid organ or stem cell transplant recipient, receiving any oral or parenteral immunosuppressive therapy, neutrophil count <500/mm^3, or an anticipated drop in the neutrophil count to <500/mm3
16. History of cancer excluding non-melanoma skin cancers or cancer more than 10 years ago
17. History of collagen vascular disease
18. Active TB
19. Women only - pregnant, planning on becoming pregnant within the next 2 months, breastfeeding, positive urine pregnancy test during screening or within 24 hours of first dose of study drug.
20. Screening laboratory tests greater than upper normal limit (ULN) or less than lower normal limit (LLN):

    1. WBCs < LLN or > ULN
    2. Neutrophils < 1500/µl (1.5 x109/L)
    3. Platelets < 100 x 10³/µl (100 x 109/L)
    4. Haemoglobin < 9.0 g/dl (90 g/L)

    f. GFR of > 40 mL/minute g. AST > 3 x upper limit of normal h. ALT > 3 x upper limit of normal i. Total Bilirubin > 1.5 x upper limit of normal
21. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer participating in the study or would make it unlikely the volunteer could complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by incidence of adverse advents | day-0 to day-28
  Occurrence of adverse events defined as a Grade II-IV toxicity (FDA's Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Subjects Enrolled in Preventative Vaccine Clinical Trials, September 2007), that are possibly or probably related to administration of SBD111

SECONDARY OUTCOMES:
Gastrointestinal Tolerability as assessed by Gastrointestinal Tolerability Questionnaire | day-0 to day-28
  Occurrence of gastrointestinal intolerability symptoms defined as a Grade II-IV toxicity

OTHER OUTCOMES:
Composition and function of the gut microbiome and presence of SBD111 in stool specimens by shotgun metagenomic sequencing | Day-0 to Day-28 and Day-56 (washout)

CONTACTS AND LOCATIONS:
Locations (1):
- Hinda and Arthur Marcus Institute for Aging Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided